CLINICAL TRIAL: NCT02985710
Title: Assessment of Small Fiber Neuropathy in Rare Diseases Using Sudoscan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amel Karaa, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P000205
Record Dates: First submitted 2016-09-12; First posted 2016-12-07 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Small Fiber Neuropathy; Fabry Disease; Ehlers Danlos Syndrome; Mitochondrial Disease
MeSH Terms: conditions — Small Fiber Neuropathy; Fabry Disease; Ehlers-Danlos Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sudoscan only (Other): Patients in this arm will only undergoing testing with Sudoscan.
  Interventions: Device: Sudoscan
- Sudoscan Plus (Other): Patients in this arm will get Sudoscan testing as well as a skin biopsy and QSART testing.
  Interventions: Device: Sudoscan; Procedure: Skin biopsy; Procedure: QSART

INTERVENTIONS:
Device: Sudoscan — The Sudoscan is a non invasive procedure and similar to standing on a scale to be weighed. Sudoscan measurements are made in compliance with the manufacturer's recommended procedures. The measurement is rapid and non-invasive, and requires no advance preparation.
Procedure: Skin biopsy — For subjects that give additional consent, skin biopsy will be done in standard fashion under sterile conditions. Assessment of nerve fiber density typically involves a 3-mm punch biopsy of skin from the leg (10 cm above the external malleolus).
  Arms: Sudoscan Plus
Procedure: QSART — QSRT (quantitative sudomotor axon reflex test) testing involves having a technician wipe the subject's arms and leg with alcohol, then tissue to wipe it dry. Electrodes filled with acetylcholine are put on three areas of the leg and one on the wrist, stimulators are turned on and sweat responses are measured.
  Other Names: Quantitative Sudomotor Autonomic Reflex Testing
  Arms: Sudoscan Plus

SUMMARY:
Sudoscan™ (Impeto Medical, Paris France) uses electrochemical skin conductance as a novel noninvasive method to detect sudomotor dysfunction. Several small studies have recently shown that Sudoscan use in the assessment of small fiber polyneuropathy (in diabetes mellitus) can be performed non-invasively, quickly and effectively. The investigators aim to study the use of Sudoscan in rare disease condition associated with small fiber polyneuropathy.

DETAILED DESCRIPTION:
Small fiber polyneuropathy (SFPN) is diagnosed through a combination of symptoms, signs and confirmatory diagnostic testing. Nerve conduction studies are not sensitive enough in most of the cases leaving the ankle skin biopsy with measurement of intraepidermal nerve fiber density (IENFD) as the main diagnostic tool. Despite its utility and reproducibility, skin biopsy is invasive, expensive and requires a central laboratory for processing and interpretation. Quantitative sudomotor axon reflex testing (QSART) is also routinely used for evaluation of small fiber neuropathy as sudomotor axons can also be involved. This test however remains technically challenging and requires testing conditions in specialized labs that are not always suitable for all patients' population. By comparing findings on skin biopsy and/or QSRT, accepted gold standard for diagnosing SFPN, the investigators seek to find faster, less-invasive ways to diagnose and monitor small-fiber polyneuropathy in rare diseases using Sudoscan measurement.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with confirmed disease: Fabry (by GLA enzymes and/or DNA testing) naïve and on ERT, Mitochondrial diseases (electron transport chain and/or DNA testing) or connective tissue diseases (clinical criteria and/or DNA testing when available)
* Consenting adults (18 years and older) who agrees and consents to skin biopsy and QSART procedure

Exclusion Criteria:

* Subjects with cognitive, psychiatric, or other problems that preclude informed consent.
* Patients with history of glucose intolerance or diabetes.
* Patient on chemotherapy
* People with any open or bleeding wounds at any sensor plate contact surface location
* People with any type of implantable device
* People with missing hand(s) and/or leg(s)
* Pregnant women or women who are uncertain about a possible pregnancy
* Patients sensitive to chemicals used to induce sweating
* Patients with heat intolerance
* Patients with bleeding disorders
* Patients on current anticoagulant therapy
* Patients with keloids on the intended biopsy site
* People with hypersensitivity to local amide-type anesthetics

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12-22 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amel Karaa, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Scientific publication at the end of the study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sudoscan Only | Sudoscan Plus
Started | 69 | 33
Completed | 65 | 33
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sudoscan Only | Sudoscan Plus | Total
Number analyzed (Participants) | 65 | 33 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 0 | 9
  Between 18 and 65 years | 50 | 27 | 77
  >=65 years | 6 | 6 | 12
Age, Continuous [Median (Standard Deviation); unit: years] | 42.4 (17.02) | 43.6 (15.35) | 42.5 (16.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 22 | 67
  Male | 20 | 11 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 33 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 33 | 98
Small fiber polyneuropathy questionnaire [Count of Participants; unit: Participants] — The SFPN questionnaire has a one week recall period and is composed of 5 domains: Miscellaneous (10 questions), Sensation (8 questions), Circulation (6 questions), Gastrointestinal (6 questions), Pelvic (4 questions) as well as a pain rating scale and clinical questions. Participants who specifically agreed to respond to the SFPN questionnaire are included and the numbers reported represent the number of participants who have responded to the questionnaire.
  Participants | 51 | 20 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Abnormal Electrochemical Skin Conductance in the Different Study Groups Who Have Clinical Symptoms Consistent With Small Fiber Polyneuropathy.
Description: The internal software of the Sudoscan will allow analysis of skin conductance in all patients and quantification into normal or abnormal. Correlation of an abnormal conductance measurement with clinical symptoms and signs of small fiber neuropathy will be evaluated for accuracy of Sudoscan measurements
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sudoscan Only | Sudoscan Plus
Number analyzed (Participants) | 65 | 33
Participants | 42 | 12

2. Secondary Outcome: Number of Patients in Whom a Specific Skin Conductance (ESC) Signature Pattern Was Detected in the Hands and/or Feet on Sudoscan Measurements.
Description: Distribution of the electrochemical skin conductance (ESC) in both hands and feet was reviewed as an indirect measure of the subject's capacity to sweat. Normative scales of adult sweat function are preloaded in the device and compared to actual measurements to determine if a subject's sweat response is reduced, which is associated with neuropathy. A positive outcome is the identification of a lower ESC in either hands or feet that distinguishes Fabry disease from other disorders and would be a reflection of the presence of SFPN.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sudoscan Only | Sudoscan Plus
Number analyzed (Participants) | 65 | 33
Participants | 21 | 16

ADVERSE EVENTS:
Time Frame: 4 years
Description: This study did not include any intervention that would cause mortality or any serious adverse events.
Arm/Group | Sudoscan Only | Sudoscan Plus
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/33
Other Adverse Events (participants affected / at risk) | 0/65 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02985710/Prot_SAP_000.pdf